CLINICAL TRIAL: NCT01058681
Title: Impacts of Metabolic Variation on the Activity of Neuroendocrine Reproductive Axis in Healthy Volunteers
Brief Title: Impacts of Metabolic Variation on Neuroendocrine Control of Reproduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Prof. François Pralong, CHUV
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Swiss national science fund; Grant number 320030-124886 (Other Grant/Funding Number: Swiss national science fund)
Record Dates: First submitted 2010-01-28; First posted 2010-01-29 (Estimated); Last update posted 2011-08-03 (Estimated); Status verified 2010-10

CONDITIONS: Neuroendocrine Reproductive Status
Keywords: LH pulsatility; GnRH regulation; isocaloric nutrition; hypercaloric nutrition; euglycemic clamps; hyperinsulinemic clamps; testosterone; LH; leptine; ghrelin; PYY; CCK; GLP-1; GIP; cortisol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- isocaloric (Other): impacts of isocaloric nutrition on LH pulsatility in euglycemic and hyperinsulinemic clamps
  Interventions: Dietary Supplement: effect of metabolic variations on LH pulsatility
- hypercaloric (Other): impacts of hypercaloric nutrition on LH pulsatility in euglycemic and hyperinsulinemic clamps
  Interventions: Dietary Supplement: effect of metabolic variations on LH pulsatility
- per os and IV glucose during the clamp (Other): impacts of per os glucose on LH pulsatility in euglycemic and hyperinsulinemic clamps
  Interventions: Dietary Supplement: effect of metabolic variations on LH pulsatility

INTERVENTIONS:
Dietary Supplement: effect of metabolic variations on LH pulsatility — Isocaloric diet: 1,5 times basal metabolism. Constitution:55% carbohydrates, 15% proteins and 30% fat.
  Hypercaloric diet: addition of 30% fat and 3 g of fructose/kg of weight to isocaloric diet.
  PO and IV glucose during clamps: PO administration of 90 mg/kg glucose at 90 minutes intervals during the clamp, and adjustment of the IV perfusion to keep euglycemia.

SUMMARY:
This study will evaluate the potential effects of a changing metabolic environment on GnRH hypothalamic neurons, by performing studies of LH pulsatility (basal and during clamp studies) in different groups of male subjects fed isocaloric and hypercaloric diets. The participation of other gastro-intestinal tract hormones to these regulations will be systematically evaluated.

ELIGIBILITY:
Inclusion Criteria:

* male
* age between 18 and 25 years old
* no known pathology
* normal physical exam
* BMI between 20 and 25 kg/m2

Exclusion Criteria:

* history of endocrine disease
* no known infertility (no conception after 12 months of regular unprotected intercourse)
* abnormal results on the initial blood tests (CBC, fasting glucose and insulin, HbA1C, TSH, free T4, LH, FSH, inhibin B and total testosterone)

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2010-01; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Luteinizing hormone (LH) pulsatility | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: François Pralong, Principal Investigator — CHUV; Vittorio Giusti, Study Director — CHUV; Luc Tappy, Study Director — CHUV; Marie-Hélène Pesant, Study Director — CHUV
Locations (1):
- CHUVaudois, Lausanne, Switzerland

REFERENCES:
- [Derived] Pesant MH, Dwyer A, Marques Vidal P, Schneiter P, Giusti V, Tappy L, Pralong FP. The lack of effect of insulin on luteinizing hormone pulsatility in healthy male volunteers provides evidence of a sexual dimorphism in the metabolic regulation of reproductive hormones. Am J Clin Nutr. 2012 Aug;96(2):283-8. doi: 10.3945/ajcn.111.030189. Epub 2012 Jul 3. PMID 22760567